CLINICAL TRIAL: NCT00612313
Title: Pediatric MDD: Sequential Treatment With Fluoxetine and Relapse Prevention
Brief Title: Sequential Treatment of Pediatric MDD to Increase Remission and Prevent Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Graham Emslie, Professor of Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH039188-01 (NIH); R01MH039188-01 (NIH); DSIR 84-CTS; NCT00599300 (obsolete NCT alias)
Record Dates: First submitted 2008-02-07; First posted 2008-02-11 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Depression
Keywords: Major Depressive Disorder; MDD; Children; Adolescents; Antidepressant; CBT
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continued medication alone (Active Comparator): Participants will receive antidepressant treatment with fluoxetine for 30 weeks
  Interventions: Drug: Fluoxetine
- Continued medication plus CBT (Experimental): Participants will receive antidepressant treatment with fluoxetine for 30 weeks plus relapse prevention cognitive behavioral therapy for the last 24 weeks of treatment
  Interventions: Drug: Fluoxetine; Behavioral: Relapse prevention cognitive behavioral therapy (CBT)

INTERVENTIONS:
Drug: Fluoxetine — Participants will take 10 to 40 mg per day of fluoxetine for 30 weeks.
  Other Names: Prozac
Behavioral: Relapse prevention cognitive behavioral therapy (CBT) — After the first 6 weeks of treatment with fluoxetine, some participants will be assigned to additionally receive relapse prevention CBT for the remaining 24 weeks of treatment. These participants will attend 10 to 12 CBT sessions, during which they will learn specific skills to reduce and prevent the occurrence of residual depressive symptoms.
  Other Names: CBT
  Arms: Continued medication plus CBT

SUMMARY:
This study will compare the effectiveness of fluoxetine alone with the effectiveness of fluoxetine with cognitive behavioral therapy in increasing recovery and preventing relapse in youth with major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a serious psychiatric disorder that affects approximately 1 out of every 12 to 15 children and adolescents. Depression can cause problems with school, family, and friends, and if left untreated, these difficulties can persist into adulthood. Treatments using antidepressants and forms of psychotherapy have been shown to be effective in reducing symptoms of depression. However, many youth experience a return of depressive symptoms within 1 to 2 years of remission. Recent studies have shown that adding cognitive behavioral therapy (CBT), a form of psychotherapy that focuses on behavioral modification, to initial antidepressant treatment may increase remission and reduce relapse rates. This study will compare the effectiveness of fluoxetine alone versus fluoxetine plus added CBT in increasing recovery and preventing relapse in youth with MDD.

Participation in this study will last 78 weeks. Potential participants will undergo initial screening, which will include interviews and questionnaires about mood, behavior, and medical history; vital sign measurements; a meeting with a psychiatrist; and lab draws and/or urine drug or pregnancy tests if indicated by the psychiatrist. All eligible participants will then begin 6 weeks of treatment with fluoxetine. During this 6-week period, participants will attend weekly study visits, which will include vital sign measurements, questionnaires on symptoms and mood, and medication dosage adjustments. At Week 6, participants will be evaluated by an independent evaluator who will determine whether their depression has significantly improved. Participants who have not improved with fluoxetine will end their study participation and will be provided with recommendations for other treatment options.

All participants who have shown significant improvement will continue to receive fluoxetine for another 24 weeks, for a total of 30 weeks of treatment. Half of these participants will be randomly assigned to additionally receive CBT for the remaining 24 weeks. All participants will attend study visits that will occur every other week for 3 months and then monthly for 3 months. These visits will last 20 to 30 minutes and will include vital sign measurements and questions about mood and behavior. Participants receiving CBT will also attend 10 to 12 CBT sessions, which will last 50 minutes each and will occur weekly for the first 4 weeks, every other week for 1.5 months, and monthly for the last 3 months. The CBT sessions will involve both individual child and parent-child sessions, which will focus on modifying depressive thoughts, feelings, and behaviors. Participants will undergo repeat evaluations with the independent evaluator at Weeks 12, 18, 24, 30, 52, and 78.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of nonpsychotic MDD (single or recurrent) for at least 4 weeks before study entry
* In good general medical health
* Normal intelligence

Exclusion Criteria:

* Lifetime history of any psychotic disorder, including psychotic depression
* Lifetime history of bipolar I and II disorders
* Alcohol or substance dependence within the 6 months before study entry
* Anorexia nervosa or bulimia within the 6 months before study entry
* Pregnant or breastfeeding females, or sexually active females not using medically acceptable means of birth control (e.g., IUD, birth control pills, barrier devices)
* Chronic medical illness (medically unstable and requires regular medication that may interfere with treatment interventions)
* Concurrent medication(s) with psychotropic effects (e.g., anticonvulsants, steroids, etc.) other than stable ADHD medication
* First degree relatives with bipolar I disorder
* Severe suicidal ideation or previous history of serious suicide attempt within this episode
* Prior failure to respond to an adequate treatment with fluoxetine (defined as at least 40 mg/day for 4 weeks)
* Non-English speaking

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham J. Emslie, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Beth D. Kennard, PsyD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- Children's Medical Center of Dallas, Outpatient Psychiatry Clinic, Dallas, Texas, United States

REFERENCES:
- [Result] Kennard BD, Emslie GJ, Mayes TL, Nakonezny PA, Jones JM, Foxwell AA, King J. Sequential treatment with fluoxetine and relapse--prevention CBT to improve outcomes in pediatric depression. Am J Psychiatry. 2014 Oct;171(10):1083-90. doi: 10.1176/appi.ajp.2014.13111460. PMID 24935082
- [Derived] Croarkin PE, Nakonezny PA, Morris DW, Rush AJ, Kennard BD, Emslie GJ. Performance and Psychometric Properties of Novel Brief Assessments for Depression in Children and Adolescents. JAACAP Open. 2024 May 27;3(2):335-343. doi: 10.1016/j.jaacop.2024.05.002. eCollection 2025 Jun. PMID 40520979
- [Derived] Emslie GJ, Kennard BD, Mayes TL, Nakonezny PA, Moore J, Jones JM, Foxwell AA, King J. Continued Effectiveness of Relapse Prevention Cognitive-Behavioral Therapy Following Fluoxetine Treatment in Youth With Major Depressive Disorder. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):991-8. doi: 10.1016/j.jaac.2015.09.014. Epub 2015 Oct 8. PMID 26598474
- [Derived] Croarkin PE, Nakonezny PA, Husain MM, Port JD, Melton T, Kennard BD, Emslie GJ, Kozel FA, Daskalakis ZJ. Evidence for pretreatment LICI deficits among depressed children and adolescents with nonresponse to fluoxetine. Brain Stimul. 2014 Mar-Apr;7(2):243-51. doi: 10.1016/j.brs.2013.11.006. Epub 2013 Dec 3. PMID 24360599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 participants began acute phase open-label treatment with fluoxetine. Of these, 144 entered the randomized control study. Results data presented are for 144 participants randomized.
Groups:
- Continued Medication Alone: n=69 Participants will receive antidepressant treatment with fluoxetine for 30 weeks
  Fluoxetine: Participants will take 10 to 40 mg per day of fluoxetine for 30 weeks.
- Continued Medication Plus CBT: n=75 Participants will receive antidepressant treatment with fluoxetine for 30 weeks plus relapse prevention cognitive behavioral therapy for the last 24 weeks of treatment
  Fluoxetine: Participants will take 10 to 40 mg per day of fluoxetine for 30 weeks.
  Relapse prevention cognitive behavioral therapy (CBT): After the first 6 weeks of treatment with fluoxetine, some participants will be assigned to additionally receive relapse prevention CBT for the remaining 24 weeks of treatment. These participants will attend 10 to 12 CBT sessions, during which they will learn specific skills to reduce and prevent the occurrence of residual depressive symptoms.
Period: Overall Study
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT
Started | 69 | 75
Completed | 52 | 62
Not Completed | 17 | 13
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lost to Follow-up | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Continued Medication Alone: Participants received antidepressant treatment with fluoxetine for 30 weeks
  Fluoxetine: Participants will take 10 to 40 mg per day of fluoxetine for 30 weeks.
- Continued Medication Plus CBT: Participants received antidepressant treatment with fluoxetine for 30 weeks plus relapse prevention cognitive behavioral therapy for the last 24 weeks of treatment
  Fluoxetine: Participants will take 10 to 40 mg per day of fluoxetine for 30 weeks.
  Relapse prevention cognitive behavioral therapy (CBT): After the first 6 weeks of treatment with fluoxetine, these participants were assigned to additionally receive relapse prevention CBT for the remaining 24 weeks of treatment. These participants attended 10 to 12 CBT sessions, during which they will learn specific skills to reduce and prevent the occurrence of residual depressive symptoms.
- Total: Total of all reporting groups
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT | Total
Number analyzed (Participants) | 69 | 75 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.2 (2.4) | 13.5 (2.7) | 13.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 30 | 37 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 23 | 43
  Not Hispanic or Latino | 49 | 52 | 101
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 54 | 64 | 118
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 69 | 75 | 144
Baseline CDRS-R [Mean (Standard Deviation); unit: units on a scale] — Childhood Depression Rating Scale - Revised (CDRS-R) Total score range: 17-113
  Scoring thresholds:
  >=40: moderate to severe depression; <=28: remission
  units on a scale | 59.2 (7.0) | 56.8 (7.1) | 58.0 (7.2)
Baseline CGI Severity [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression - Severity Range: 1-7
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severly ill
  7. Among the most extremely ill patients
  units on a scale | 5.3 (0.69) | 5.1 (0.7) | 5.2 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Time to Remission
Description: Remission is defined as CDRS-R <=28. Timing of remission is based on clinical assessment using the CDRS-R and K-Life to identify the week at which point the patient remitted.
Time Frame: 30 weeks
Measure: Mean (Standard Error); unit: weeks
Groups:
- Continued Medication Alone: Participants received antidepressant treatment with fluoxetine for 30 weeks
  Fluoxetine: Participants took 10 to 40 mg per day of fluoxetine for 30 weeks.
- Continued Medication Plus CBT: Participants received antidepressant treatment with fluoxetine for 30 weeks plus relapse prevention cognitive behavioral therapy for the last 24 weeks of treatment
  Fluoxetine: Participants took 10 to 40 mg per day of fluoxetine for 30 weeks.
  Relapse prevention cognitive behavioral therapy (CBT): After the first 6 weeks of treatment with fluoxetine, these participants were assigned to additionally receive relapse prevention CBT for the remaining 24 weeks of treatment. These participants will attend 10 to 12 CBT sessions, during which they learned specific skills to reduce and prevent the occurrence of residual depressive symptoms.
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT
Number analyzed (Participants) | 69 | 75
weeks | 13.67 (1.17) | 11.33 (0.95)

2. Primary Outcome: Relapse
Description: Relapse was defined as:
  1) CDRS-R score >=40 with a history of 2 weeks of clinical deterioration or 2) CDRS-R<40, but with a 2 week history of significant clinical deterioration.
Time Frame: Measured at Weeks 12, 18, 24, and 30
Population: Only participants who achieved remission were analyzed for relapse rates, as only remitted patients can experience a relapse of depression.
Measure: Number; unit: probability of relapse (%)
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT
Number analyzed (Participants) | 52 | 64
probability of relapse (%)
  Week 12 | 3 | 1
  Week 18 | 10 | 3.5
  Week 24 | 20.5 | 7
  Week 30 | 26.5 | 9

3. Secondary Outcome: K-Life (Time Well)
Description: K-Life interview was conducted at Weeks 6, 12, 18, 24, and 30, with ratings for depressive illness for each week throughout the study.
  Ratings definitions: 1=Normal, no residual symptoms; 2=Presence of 1 or more symptosm in no more than mild degree; 3=Considerably less psychopathology than full criteria, but still obvious evidence of disorder with no more than moderate impairment; 4=Does not meet full criteria, but has major symptoms or impairment from the disorder; 5=Meets full criteria, but no extreme impairment; 6=Meets full criteria, and either has prominent psychotic symptoms or extreme impairment.
  Time well is defined as each week the depression rating was a 1 or 2. Percent time well was defined as each week the depression rating was a 1 or 2 divided by the total number of weeks in the study.
  Statistic: anova
Time Frame: 30 weeks
Measure: Mean (Standard Deviation); unit: Weeks spent well
Groups:
- Continued Medication Alone: Participants received antidepressant treatment with fluoxetine for 30 weeks
  Fluoxetine: Participants took 10 to 40 mg per day of fluoxetine for 30 weeks.
  n=69
- Continued Medication Plus CBT: Participants received antidepressant treatment with fluoxetine for 30 weeks plus relapse prevention cognitive behavioral therapy for the last 24 weeks of treatment
  Fluoxetine: Participants took 10 to 40 mg per day of fluoxetine for 30 weeks.
  Relapse prevention cognitive behavioral therapy (CBT): After the first 6 weeks of treatment with fluoxetine, these participants were assigned to additionally receive relapse prevention CBT for the remaining 24 weeks of treatment. These participants will attend 10 to 12 CBT sessions, during which they learned specific skills to reduce and prevent the occurrence of residual depressive symptoms.
  n=75
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT
Number analyzed (Participants) | 69 | 75
Weeks spent well | 12.8 (9.5) | 16.0 (9.1)
Statistical Analysis 1: Comparison: Continued Medication Alone vs Continued Medication Plus CBT; Test type: Superiority or Other; p = .02, Regression, Poisson — The estimated rate of time spent well was evaluated using a Poisson regression with adjustment for CDRS-R score at the end of the acute phase, age group, and gender; Difference in percentages = 9.7 — Differencein percentages represents estimated percentage for medication management + CBT Arm minus estimated percentage for medication management only Arm

4. Secondary Outcome: Remission
Description: Remission is defined as CDRS-R <=28 (up through week 30) or at least 8 consecutive weeks of a K-Life rating of 1 or 2. Timing of remission is based on clinical assessment using the CDRS-R and K-Life to identify the week at which point the patient remitted.
Time Frame: Weeks 52 and 78
Measure: Number; unit: Probability of remission (%)
Groups:
- Continued Medication Alone: Participants received antidepressant treatment with fluoxetine for 30 weeks
  Fluoxetine: Participants took 10 to 40 mg per day of fluoxetine for 30 weeks.
  Treatment was uncontrolled after week 30.
- Continued Medication Plus CBT: Participants received antidepressant treatment with fluoxetine for 30 weeks plus relapse prevention cognitive behavioral therapy for the last 24 weeks of treatment
  Fluoxetine: Participants took 10 to 40 mg per day of fluoxetine for 30 weeks.
  Relapse prevention cognitive behavioral therapy (CBT): After the first 6 weeks of treatment with fluoxetine, these participants were assigned to additionally receive relapse prevention CBT for the remaining 24 weeks of treatment. These participants will attend 10 to 12 CBT sessions, during which they learned specific skills to reduce and prevent the occurrence of residual depressive symptoms.
  Treatment was uncontrolled after week 30.
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT
Number analyzed (Participants) | 69 | 75
Probability of remission (%)
  Week 52 | 89 | 94
  Week 78 | 92 | 96

5. Secondary Outcome: Relapse
Description: Up through week 30, relapse was defined as:
  1) CDRS-R score >=40 with a history of 2 weeks of clinical deterioration or 2) CDRS-R<40, but with a 2 week history of significant clinical deterioration.
  From week 31-78, relapse was assessed using the K-Life. Relapse was defined as at least 2 weeks of a K-Life rating of 5 or 6; participants may also be identified as relapsing with a K-Life rating of 4 if the rating was for several weeks and not strictly related to stressful life events.
Time Frame: Weeks 52 and 78
Population: as for outcome 2
Measure: Number; unit: Probability of Relapse (%)
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT
Number analyzed (Participants) | 54 | 67
Probability of Relapse (%)
  Week 52 | 49 | 27
  Week 78 | 62 | 36

6. Primary Outcome: Remission
Description: Remission is defined as CDRS-R <=28.
Time Frame: Measured at Weeks 12, 18, 24, and 30
Measure: Number; unit: probability of remitting (%)
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT
Number analyzed (Participants) | 69 | 75
probability of remitting (%)
  Week 12 | 59 | 68
  Week 18 | 71 | 79
  Week 24 | 80 | 86
  Week 30 | 84 | 90

ADVERSE EVENTS:
Arm/Group | Continued Medication Alone | Continued Medication Plus CBT
Serious Adverse Events (participants affected / at risk) | 7/69 | 9/75
Other Adverse Events (participants affected / at risk) | 0/69 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continued Medication Alone (N=69) | Continued Medication Plus CBT (N=75)
Hospitalization for Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization for Suicidal Ideation (Psychiatric disorders) | 3 (3) | 5 (5)
Hospitalization for Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization for medical conditions (General disorders) | 2 (2) | 3 (5)
Suicidal behavior that did not result in hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
* Primary outcomes based on data through 30 weeks.
* Participants were not blinded to treatment assignment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No